CLINICAL TRIAL: NCT06378125
Title: A Phase I, Double-blind, Randomised, Placebo-controlled, Single-ascending and Multiple-ascending Dose Trial to Evaluate the Safety and Pharmacokinetics of Oral Controlled-ileal-release Nicotinic Acid (CIR-NA) Compared to Immediate-release Nicotinic Acid and Placebo in Healthy Subjects and Subjects With Prediabetes
Brief Title: Evaluation of Safety and Pharmacokinetics of Oral Controlled-ileal-release Nicotinic Acid (CIR-NA) Compared to Immediate-release Nicotinic Acid and Placebo in Healthy Subjects and Subjects With Prediabetes
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University Hospital Schleswig-Holstein (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Other
Other Study IDs: CIR-NA I
Record Dates: First submitted 2024-04-17; First posted 2024-04-22 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2024-04

CONDITIONS: Safety Issues; Pharmacokinetic
Keywords: Nicotinic Acid; Prediabetes
MeSH Terms: conditions — Prediabetic State | interventions — Sagittal Abdominal Diameter; Single Person

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Double (Participant, Investigator)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- healthy subjects healthy subjects (Experimental): single-ascending and multipleascending doses (SAD/MAD)
  Interventions: Drug: controlled-ileal-release nicotinic acid (SAD/ MAD/MD) single- and multiple-ascending dose (SAD/MAD) or multiple dose (MD); Drug: immediate-release nicotinic acid (SAD); Drug: Placebo controlled-ileal-release nicotinic acid (SAD/MAD); Drug: Placebo immediate-release nicotinic acid (SAD)
- subjects with prediabetes (Experimental): multiple dose (MD)
  Interventions: Drug: controlled-ileal-release nicotinic acid (SAD/ MAD/MD) single- and multiple-ascending dose (SAD/MAD) or multiple dose (MD)

INTERVENTIONS:
Drug: controlled-ileal-release nicotinic acid (SAD/ MAD/MD) single- and multiple-ascending dose (SAD/MAD) or multiple dose (MD) — A double-blind, randomised, placebo-controlled, single-ascending and multiple-ascending dose trial to evaluate the safety and pharmacokinetics of oral controlled-ileal-release nicotinic acid (CIR-NA) compared to immediate-release nicotinic acid and placebo in healthy subjects and subjects with prediabetes.
  Other Names: CIR-NA (SAD/MAD/MD)
Drug: immediate-release nicotinic acid (SAD) — A double-blind, randomised, placebo-controlled, single-ascending and multiple-ascending dose trial to evaluate the safety and pharmacokinetics of oral controlled-ileal-release nicotinic acid (CIR-NA) compared to immediate-release nicotinic acid and placebo in healthy subjects and subjects with prediabetes.
  Other Names: ImR-NA (SAD)
  Arms: healthy subjects healthy subjects
Drug: Placebo controlled-ileal-release nicotinic acid (SAD/MAD) — A double-blind, randomised, placebo-controlled, single-ascending and multiple-ascending dose trial to evaluate the safety and pharmacokinetics of oral controlled-ileal-release nicotinic acid (CIR-NA) compared to immediate-release nicotinic acid and placebo in healthy subjects and subjects with prediabetes.
  Other Names: no active substance (SAD/MAD)
  Arms: healthy subjects healthy subjects
Drug: Placebo immediate-release nicotinic acid (SAD) — A double-blind, randomised, placebo-controlled, single-ascending and multiple-ascending dose trial to evaluate the safety and pharmacokinetics of oral controlled-ileal-release nicotinic acid (CIR-NA) compared to immediate-release nicotinic acid and placebo in healthy subjects and subjects with prediabetes.
  Other Names: no active substance (SAD)
  Arms: healthy subjects healthy subjects

SUMMARY:
A double-blind, randomised, placebo-controlled, single-ascending and multiple-ascending dose trial to evaluate the safety and pharmacokinetics of oral controlled-ileal-release nicotinic acid (CIR-NA) compared to immediate-release nicotinic acid and placebo in healthy subjects and subjects with prediabetes.

DETAILED DESCRIPTION:
Recently, administration of one form of vitamin B3, Nicotinamide (NAM), has been shown to improve the host-microbiome interaction in a mouse model, especially when administered in a controlled-release formulation targeting the ileocolic region. Thus, NAM and also the other form of vitamin B3, Nicotinicacid (NA), were identified as promising candidates for a gut-targeted microbiome intervention.

As the upper gastrointestinal tract efficiently absorbs amino acids and vitamins, simply increasing the NA and/or NAM content in human food would not be expected to deliver these molecules in sufficient amounts into the lower ileum and colon, where most of the microbiota are located. Moreover, adverse effects such as flushing or gastrointestinal symptoms can occur under high and immediately systemically available dosage of NA. Therefore, the novel CIR-NA formulation will be applied to deliver NA to the lower ileum and colon to tar-get the gut microbiome, while largely avoiding systemic exposure, as the terminal ileum and colon have a much lower absorptive capacity than the stomach and upper small intestine.

Both in the single- and multiple-ascending (SAD/MAD) part of the study, CIR-NA or placebo tablets will be self-administered orally, with daily doses of 100 mg (1 tablet), 200 mg (2 tablets), 500 mg (5 tablets) or 1,000 mg CIR-NA (10 tablets) or the corresponding amounts of placebo tablets. In the SAD part, an additional dose of 2,000 mg CIR-NA or placebo (20 tablets) will be self-administered.After completion of the SAD and the 200 mg MAD part in healthy subjects, an additional mul-tiple dose part (200 mg/d CIR-NA) in subjects with PreD (MD-PreD part) will start in parallel to the further dose groups of the MAD part.

ELIGIBILITY:
Main inclusion and exclusion criteria

Inclusion criteria for the SAD and MAD parts with healthy subjects:

1. Male and female subjects aged 18 to 65 years.
2. Healthy subjects without relevant medical conditions.
3. Ability to understand and comply with the protocol.
4. Signed written Informed Consent.
5. A BMI of 18.5 to 29.99 kg/m².
6. Non-smoker or light smoker (average of <7 cigarettes per week) and no history of longterm, heavy smoking (>10 pack-years).

Inclusion criteria for the MD-Part (subjects with prediabetes):

1. Male and female subjects aged 18 to 65 years.
2. Previously diagnosed prediabetes with confirmation via the HbA1c level (5.7 to < 6.5%) at the screening visit.
3. Subjects without relevant medical conditions and without clinically significant impairment of renal or hepatic function.
4. Ability to understand and comply with the protocol.
5. Signed written Informed Consent.
6. A body mass index of 25 to 40 kg/m², both inclusive .
7. Non-smoker or light smoker (average of <7 cigarettes per week) and no history of longterm, heavy smoking (>10 pack-years).

Exclusion criteria for the SAD, MAD and MD part with healthy subjects and subjects with prediabetes:

1. Pre-existing relevant medical conditions.
2. Clinically relevant abnormal findings in medical history or screening assessments.
3. Participation in a clinical study.
4. Use of any prescribed or over-the-counter medication, food supplements or herbal preparations.
5. Use of antibiotics (systemic or gut-acting [non-absorbed]).
6. Pregnant or breastfeeding women or women of childbearing potential and male participants with female partners of childbearing age not using highly effective contraception till at least 1 month after last dosing of investigational medicinal product (IMP).
7. Legal incapacity.
8. Indications that the patient may be unable to comply with the study procedures, e.g. language barriers precluding adequate understanding or cooperation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-12-19 (Actual); Primary Completion 2024-11-12 (Actual); Study Completion 2024-11-12 (Actual)

PRIMARY OUTCOMES:
Treatment-Emergent Adverse Events [Safety and Tolerability] | up to 60 days
  Adverse Events (AEs) during treatment period
Treatment-Emergent Serious Adverse Events [Safety and Tolerability] | up to 60 days
  Serious Adverse Events (SAEs) during treatment period
Haemoglobin | up to 60 days
  Haemoglobin (Hb) in %
White blood cells | up to 60 days
  White blood cell (WBC) count as x10^9/l
Blood creatinine | up to 60 days
  Blood Creatinine in mmol/L
Blood urea | up to 60 days
  Urea in mmol/L
Blood uric acid | up to 60 days
  Uric acid in mmol/L
Glomerular filtration rate | up to 60 days
  Glomerular filtration rate (GFR, automatically calculated by the laboratory based on creatinine values) GFR in ml/min/1.73m2
Blood ALT | up to 60 days
  Alanine transaminase (ALT) in U/l
Blood AST | up to 60 days
  Aspartate transaminase (AST) in U/l
Blood GGT | up to 60 days
  Gamma glutamyl transferase (GGT) in U/l

CONTACTS AND LOCATIONS:
Overall Officials: Susanna Nikolaus, Prof. Dr., Principal Investigator — University Medical Center Schleswig-Holstein, Campus Kiel
Locations (1):
- University Medical Center Schleswig-Holstein, Campus Kiel, Kiel, Schleswig-Holstein, Germany

IPD SHARING:
Plan to Share IPD: No